CLINICAL TRIAL: NCT00272623
Title: A Prospective, Randomized Trial Comparing Seldinger Technique Versus Venous Cut-Down for Placement of Totally Implantable Venous Access Ports
Brief Title: Seldinger Technique Versus Venous Cut-Down for Placement of Totally Implantable Venous Access Ports
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: StV 33-2005
Record Dates: First submitted 2006-01-03; First posted 2006-01-06 (Estimated); Last update posted 2009-06-03 (Estimated); Status verified 2009-06

CONDITIONS: Catheters, Indwelling
Keywords: Catheter, Indwelling; Indwelling Catheter; Indwelling Catheters; Implantable Catheters; Catheter, Implantable; Catheters, Implantable; Implantable Catheter; In-Dwelling Catheters; Catheter, In-Dwelling; Catheters, In-Dwelling; In Dwelling Catheters; In-Dwelling Catheter; Venous Reservoirs; Reservoir, Venous; Reservoirs, Venous; Venous Reservoir; Vascular Access Ports; Access Port, Vascular; Access Ports, Vascular; Port, Vascular Access; Ports, Vascular Access; Vascular Access Port

INTERVENTIONS:
Procedure: Seldinger technique or venous cut-down for port placement

SUMMARY:
Since the first placement of a totally implantable venous access port (TIVAP) by Niederhuber et al in 1982 its application to provide long-term central venous access has dramatically increased. These systems have dramatically simplified the administration of chemotherapy and parenteral nutrition as well as the repetitive collection of blood samples.

Initial retrospective studies have focused on the complications associated with different implantation techniques. Subsequently, major attention has been payed to the comparison of distinct types of TIVAPs. To date a variety of approved port systems are available. These devices can be either implanted using the Seldinger technique or by venous cut-down of the cephalic vein Despite the global use of these established implantation procedures prospective, randomized trials directly comparing these two approaches are still lacking. So, the choice, which technique to use is left to the surgeon's preference.

The aim of this study is to directly compare the Seldinger technique versus cephalic vein cut down for placement of TIVAPs in respect of implantation success rate, operation time and perioperative morbidity.

DETAILED DESCRIPTION:
Since the first placement of a totally implantable venous access port (TIVAP) by Niederhuber et al in 1982 its application to provide long-term central venous access has dramatically increased. These systems have dramatically simplified the administration of chemotherapy and parenteral nutrition as well as the repetitive collection of blood samples.

Initial retrospective studies have focused on the complications associated with different implantation techniques. Subsequently, major attention has been payed to the comparison of distinct types of TIVAPs. To date a variety of approved port systems are available. These devices can be either implanted using the Seldinger technique or by venous cut-down of the cephalic vein Despite the global use of these established implantation procedures prospective, randomized trials directly comparing these two approaches are still lacking. So, the choice, which technique to use is left to the surgeon's preference.

The aim of this study is to directly compare the Seldinger technique versus cephalic vein cut down for placement of TIVAPs in respect of implantation success rate, operation time and perioperative morbidity.

After an informed consent has been obtained, patients will be randomized as follows: By means of sealed envelopes a total of 152 patients will be allocated either to TIVAP placement using Seldinger technique or by venous cut down (n= 76 in each group).

Operations will be performed in local or general anaesthesia either on an outpatient basis or via 24h-admission. Changes of technique due to catheter implantation failure, operation time and intraoperative complications will be assessed during the procedure. Postoperative examination will be standardized in both groups, i.e. chest radiography (to confirm catheter placement and to exclude pneumothorax) as well as final clinical examination at discharge or before patient transfer.

ELIGIBILITY:
Inclusion Criteria:

* Oncological patients with an indication for a long-term parenteral treatment
* Age > 18 years
* Elective operations only

Exclusion Criteria:

* Patients with limited German proficiency (informed consent not possible)
* Anticoagulation (INR >2.5), coagulopathy, Tc<60'000/mI
* Bilateral intervention/irradiation on shoulder, clavicle or breast

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2006-01; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Implantation success rate

SECONDARY OUTCOMES:
Amount of puncture attempts needed (new perforation of the skin)
Intraoperative change of surgical technique
Operation time
Intra-/perioperative complications (arterial puncture, major arrhythmia, pneumothorax, haemorrhage/haematoma)

CONTACTS AND LOCATIONS:
Overall Officials: Markus Weber, MD, Principal Investigator — Dept. of Visceral and Transplantation Surgery, University Hospital Zurich
Locations (1):
- Dept. of Visceral and Transplantation Surgery, Zurich, Canton of Zurich, Switzerland

REFERENCES:
- [Derived] Nocito A, Wildi S, Rufibach K, Clavien PA, Weber M. Randomized clinical trial comparing venous cutdown with the Seldinger technique for placement of implantable venous access ports. Br J Surg. 2009 Oct;96(10):1129-34. doi: 10.1002/bjs.6730. PMID 19731229